CLINICAL TRIAL: NCT05956067
Title: Chromatic Retinal Stimulation to Reduce Chronic Pain and Pain Sensitivity
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Anticipate resuming after repair of our stimulus
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-1301
Record Dates: First submitted 2023-06-28; First posted 2023-07-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-01

CONDITIONS: Chronic Low-back Pain; Chronic Pain; Fibromyalgia
MeSH Terms: conditions — Chronic Pain; Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Equal energy white stimulus (Experimental): Equal energy white light at 500 lux. The International Commission on Illumination (CIE) coordinates of this light are (x=y=0.33), indicating that the stimulus appears uniformly white which means that the activation of each of the three classes of photoreceptors are equivalent, thus silencing any chromatic opponency. The stimulus will be delivered by a portable battery-operated ganzfeld light stimulation device for 2 hours per day for 5 consecutive days.
  Interventions: Device: Equal Energy White stimulation
- Green light stimulus (Experimental): Green light at 500 lux. Participants will view 545 nm green light delivered via a portable battery-operated ganzfeld light stimulation device for 2 hours per day for 5 consecutive days.
  Interventions: Device: Green Light stimulation
- S-cone modulating white light (Experimental): The S-cone modulating light stimulus will alternate between two light conditions at 500 lux that will activate the S-cones by about 100x differentially between the two conditions while maintaining the L- an M-cones at constant activation between the two alternating conditions using 427 nm versus 545 nm light. The stimulus will be delivered by a portable battery-operated ganzfeld light stimulation device for 2 hours per day for 5 consecutive days.
  Interventions: Device: S-cone modulating white light

INTERVENTIONS:
Device: Green Light stimulation — A portable battery-operated ganzfeld light display will be used to deliver green light for 2 hours per day for 5 consecutive days.
  Arms: Green light stimulus
Device: Equal Energy White stimulation — A portable battery-operated ganzfeld light display will be used to deliver white light for 2 hours per day for 5 consecutive days.
  Arms: Equal energy white stimulus
Device: S-cone modulating white light — A portable battery-operated ganzfeld light display will be used to deliver S-cone modulating light for 2 hours per day for 5 consecutive days.
  Arms: S-cone modulating white light

SUMMARY:
Participants with chronic pain conditions including chronic low back pain and fibromyalgia may benefit from light stimuli presented to the retina to reduce chronic pain severity and pain sensitivity. Participants will be recruited into this study and will be presented with one of three uniform light stimuli via a wide-field ganzfeld in three conditions to determine the retinal mechanisms that reduce pain. This work will lead to a greater understanding of retinal mechanisms that contribute to pain and will assist the design of future studies to harness the potential of light based pain therapies.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to 18 and less than or equal to 65.
* Individuals who have been diagnosed with fibromyalgia or chronic low back pain by their physician.
* Individuals who experience an average pain severity greater than 4/10 in intensity at baseline.
* Willingness to wear a battery-operated portable ganzfeld light stimulator device for 2 hours per day at the same time each day (ideally complete the light therapy session between 5 am-10 am each morning) for 5 days.
* Alert and oriented, and able to provide informed consent
* Ability to read and speak English to complete validated questionnaires.

Exclusion Criteria:

* Vision disorders or conditions resulting in severe vision impairment or blindness
* Individuals with self-report of color blindness
* Prisoner Status
* Pregnancy
* No other history or condition that would, in the investigator's judgment, indicate that the patient would very likely be non-compliant with the study or unsuitable for the study (e.g., might interfere with the study, confound interpretation, or endanger the patient).
* History of seizure disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2026-07-17 (Estimated); Study Completion 2026-07-29 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Percent follow-up | 1 week
  Percent follow-up for 1 week baseline visit. Follow-up greater than 70% will be considered feasible.
Feasibility: Percent of flash surveys completed | 1 week
  Percent of flash surveys completed during light stimulation period. 0% is the lowest and 100% is the highest. Higher percentages indicate greater percent of flash surveys completed.
Feasibility: Self-reported light stimulation sessions completed | 1 week
  Self-reported light stimulation sessions completed by flash survey administered after each light stimulation session over the 5 day stimulation period. Number of sessions will be reported the minimum is 0 and the maximum is 5.

SECONDARY OUTCOMES:
Change in pain intensity after stimulation | Baseline, 1 week
  Pain intensity measured by a 0-10 numeric rating scale for overall pain. 0 represents no pain, and 10 represents the worst pain imaginable.
Change in pressure pain threshold | Baseline, 1 week
  Pressure Pain Threshold is the threshold in which pain is experienced in response to increasing force applied to the trapezius measured by a pressure algometer in kilograms of force per square centimeter (kgf/cm^2). The higher the value, the higher the threshold. The maximum is 10 kgf/cm^2 and minimum is 0.
Change in Conditioned Pain modulation | Baseline, 1 week
  Conditioned Pain modulation magnitude will be calculated as the difference in mean pressure pain threshold (kgf/cm^2) measured prior to and during the conditioning stimulus (cold water bath), with increases in pressure pain threshold during conditioning interpreted as evidence of efficient endogenous pain inhibition.
Change in Temporal Summation | Baseline, 1 week
  Temporal Summation. The investigators will evaluate temporal summation using a 40g Neuropen applied to the skin of the volar forearm and lumbar region, following a train of 10 identical stimuli (1 Hz). Participants will report retrospectively, the pain intensity of the 1st and 10th pinprick using a 0-10 numerical rating scale (NRS). 0 is the minimum and 10 is the maximum pain intensity that will be reported.
Change in activity measured with an accelerometer | 1 week prior to baseline and 1 week during light stimulation
  Activity will be measured by an accelerometer. Average daily step count for the duration of the stimulus. Average non-sedentary time in minutes will able be determined over the stimulation period and compared to the data collected over the 1 week run-in period.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Mauck, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University Of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 18 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 1 year after completion of the study and will be available for an additional 2 years.
Access Criteria: Data use agreement with University before deidentified information requested will be shared.